CLINICAL TRIAL: NCT06452875
Title: PRIMARY NEEDLE KNIFE FISTULOTOMY FOR BILIARY CANNULATION IN A CONSECUTIVE GROUP OF PATIENTS
Brief Title: PRIMARY NEEDLE KNIFE FISTULOTOMY
Status: Completed | Type: Observational
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Luis Lopes, PhD, University of Minho
Other Study IDs: 30/2021
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pancreatitis
Keywords: ERCP; Biliary cannulation; Needle-knife fistulotomy; Standard cannulation methods
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Primary Needle Knike Fistulotomy — After verifying the eligibility of the papillary morphology (excluding flat or diverticular papillae according to Viana's classification), access to the bile duct will be initiated using the primary needle knife fistulotomy technique. After the first contact of the needle knife with the papilla, the endoscopist will have a total of 8 minutes, after which he can change to other cannulation techniques (eg standard cannulation methods through the papillary orifice) or even stop the procedure.
  During ERCP all patients will be submitted to PEP prophylaxis with indomethacin. Also as a prophylactic PEP measure a pancreatic stent will be placed whenever there is cannulation or opacification of the Wirsung duct. For the purpose of this study, a dedicated form (attached) will be created with the various variables to be analyzed.

SUMMARY:
Evaluate the outcomes of NKF as an initial method for biliary access.

DETAILED DESCRIPTION:
Introduction

A previous feasibility study has suggested that needle knife fistulotomy (NFK) as an initial method for biliary access in patients with stones is associated with high levels of success and low rate of complications. This study evaluated the outcomes of NKF as an initial method for biliary access, in a large number of patients with any type of biliary pathology (tumors and stones), on the basis of success rate, complications and factors associated with success and complications.

Financial resources

All participants included in this study will perform ERCP, laboratory tests and other complementary diagnostic tests after a duly justified medical prescription. Therefore there are no additional costs or consumption of hospital resources.

Ethical considerations

In this study, participants will be included after informed consent. Anonymity and confidentiality will be safeguarded by assigning an individual numeric code. It will also be explained the possibility of withdrawing from the study at any time, with the guarantee of the total elimination of data. All researchers involved in the study will adhere to the Rules of Ethical Conduct and Best Practices in order to comply with the precepts of the Declaration of Helsinki, the Convention on Human Rights and Biomedicine, the guidelines of the Council for International Organizations of Medical Sciences and the Guide to Good Clinical Practice.

Statistical analysis

Qualitative variables will be summarized using absolute and relative frequencies, and quantitative variables will be summarized using the mean and standard deviation or the median and interquartile range, depending on their distribution profiles. The normality of the quantitative variables will be assessed using the histogram distribution.

Relations between categorical variables will be assessed using a chi-square test and Fisher´s exact test. Differences between two or more groups of independent non-normally distributed quantitative variables will be evaluated using a Kruskal-Wallis test.

To explain the risk of pancreatitis, a binomial logistic regression model with multiple predictors will be performed.

The null hypothesis will be rejected when the test statistics p-values are less than <0.05. Statistical analysis, sample size calculation and graphics will be performed using Stata software (StataCorp. 2015. Stata Statistical Software: Release 14. College Station, StataCorp LP)

Expected results

The results of this study will contribute to a better understanding of what is the best algorithm to follow when performing an ERCP.

ELIGIBILITY:
Inclusion Criteria:

* ERCP with indication for biliary access
* Naïve papilla

Exclusion Criteria:

* Patients unable to sign or understand the informed consent
* Patients with surgically altered anatomy
* Patients with tumors of the papilla
* Previous sphincterotomy
* Spontaneous papillary fistula
* Papilla not visualized

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * ERCP with indication for biliary access
  * Naïve papilla (excluding flat or diverticular papillae according to Viana's classification)
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 30 days from the procedure
  Comparison of adverse event rate between the two strategies
Technical success | 1 day (same day of the procedure)
  Comparison of technical success between the two strategies

CONTACTS AND LOCATIONS:
Locations (1):
- ULS Nordeste, Bragança, Portugal

IPD SHARING:
Plan to Share IPD: Undecided